CLINICAL TRIAL: NCT04214405
Title: One Point Versus Two Point Fixation of Tripodal Zygomatic Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Gamal Thabet (Other)
Responsible Party: Sponsor-Investigator, Mohamed Gamal Thabet, principal investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mohamed Gamal Thabet
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Assessment of Proper Union of Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- union of fractures (Experimental): proper union of zygomatic fractures
  Interventions: Procedure: fixation of tripodal zygomatic fractures

INTERVENTIONS:
Procedure: fixation of tripodal zygomatic fractures — One point versus two point fixation of tripodal zygomatic fractures

SUMMARY:
The zygomatic bone defines the anterior and lateral projection of the face and articulates with the frontal, sphenoid,temporal, and maxillary bones. The zygomatic complex is responsible for the protection of the orbital contents and the mid-facial contour. Fracture of the zygomatic complex is one of the most common facial injuries in maxillofacial trauma and predominately appears in young adult males. The etiology of zygomatic complex fractures primarily includes road traffic accidents, violent assaults, falls and sports injuries. The main clinical features of zygomatic complex fractures include diplopia, enophthalmos, subconjunctival ecchymosis, extraocular muscle entrapment, cosmetic deformity with depression of the malar eminence, malocclusion and neurosensory disturbances of the infraorbital nerve. Diagnosis of zygomatic complex fractures is usually clinical with confirmation by computed tomography (CT) scan. Zygomatic complex fractures with no or minimal displacement are often treated without surgical intervention, whereas fractures with functional or esthetic impairments often necessitate surgical intervention. Various surgical approaches and treatment strategies have been proposed to obtain successful treatment outcome, including the Gilles temporal approach, eyebrow, upper eyelid, transconjunctival, infraciliary lower eyelid, and intraoral vestibular approaches. The surgical approach for adequate reduction of zygomatic complex fractures must ensure a good functional and cosmetic result. Surgical reduction of zygomatic fractures by an intraoral surgical approach was first described in1909 by Keen, and several studies have subsequently documented the treatment outcome after open reduction of zygomatic complex fractures by an intraoral surgical approach.

DETAILED DESCRIPTION:
This study is a prospective clinical intervention study where the admitted patients do lab investigation as CBC, coagulation profile ,Kidney function test and Imaging as CT maxillofacial with axial and coronal cuts. Patients will be assigned randomly into either one of the two groups under the study using concealed envelope. Under general anaesthesia with oral or naso-tracheal intubation, open reduction and internal fixation of tripod zygomatic fractures will be done using miniplates and screws at one point (zygomaticomaxillary area) or at two points (zygomaticomaxillary and frontozygomatic areas).

ELIGIBILITY:
Inclusion Criteria:

* (a) Adult patients with maxillofacial fractures including tripodal zygomatic fractures as determined on clinical and radiological finding (b) Isolated tripodal fracture zygoma

Exclusion Criteria:

* patients with Le Fort I/II/III fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
union of fractures | 2 months
  assessment of proper union of fractures

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Gamal, Principal Investigator — Assiut University
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Clinical Study Report — https://www.ncbi.nlm.nih.gov — Birgfeld CB, Mundinger GS, Gruss JS. Evidence-based medicine: Evaluation and treatment of zygoma fractures. Plast Reconstr Surg 2017;139(1): 168e-80e.[http://dx.doi.org/10.1097/PRS.0000000000002852] [PMID: 28027253]